CLINICAL TRIAL: NCT02430571
Title: A Prospective, Single-Center, Open Label, Within-Subject Case Series to Evaluate the Identification of Anatomical Markers in the Gastrointestinal Tract Using the KANGAROO™ Feeding Tube With IRIS Technology
Brief Title: Case Series to Evaluate the Identification of Anatomical Markers Using the KANGAROO™ Feeding Tube
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVIRIS0465
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Enteral Nutrition, Feeding Tube Placement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, single-center, open label, within-subject clinical trial to evaluate the identification of anatomical markers in the gastrointestinal tract using the IRIS feeding tube. The trial will evaluate hospitalized subjects who require short-term enteral feeding with an anticipated duration of at least 3 days while in an intensive care unit (ICU) or step-down unit. Eligible men and women at least 18 years of age who give voluntary, written informed consent to participate in the clinical investigation will be included as subjects. If a potential subject is incapacitated and unable to provide informed consent, a designated legally authorized representative will be allowed to provide the informed consent on behalf of the subject to allow their participation in the study. Study entry will be defined as the point of signed informed consent. A Prospective, Single-Center, Open Label, Within-Subject Case Series to Evaluate the Identification of Anatomical Markers in the Gastrointestinal Tract Using the KANGAROO™ Feeding Tube with IRIS Technology

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized male and female patients in a monitored setting (i.e.; ICU or Step-Down Unit) who require and are eligible for short-term enteral (nasal or oral) feeding per standard of care with an expected duration of at least 3 days.
2. The subject or a legally authorized representative is able to understand and willing to give written informed consent.
3. Be a man or woman of 18 years or older
4. Have uncomplicated naso- and oropharyngeal anatomy based upon a focused physical examination

Exclusion Criteria:

1. Women and men under the age of 18 years
2. Female patients who are known to be pregnant or lactating
3. Incarcerated or imprisoned individuals
4. Hemodynamic instability with an inability to maintain a MAP > 65 mm Hg on vasopressors
5. Patients who are currently enrolled in an investigational or interventional drug or device clinical trial
6. Patients who have been previously enrolled into this study
7. Individuals, who, in the opinion of the Principal Investigator, have any medical, social or psychological condition that would compromise their participation and follow-up in this clinical investigation
8. Known basal skull fractures
9. Unrepaired known GI perforation or leak
10. Recent adequate upper GI bleed that may obscure images
11. Esophageal varices > Grade 2
12. Subjects with known anomalies precluding gastric or intestinal insertion (via either nasally or orally)
13. Known obstruction of the gastrointestinal tract
14. Known bowel ischemia or any other contraindication for enteral feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring nasogastric feeding tube in an ICU or step-down unit
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The ability of the clinician to recognize anatomical markers in the gastrointestinal tract using the IRIS feeding tube | during the feeding tube placement procedure
  the following anatomical structures will be noted if visualized and the depth of feeding tube will also be recorded corresponding to the visualized structure: trachea/carina, esophagus, stomach

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wischmeyer, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes